CLINICAL TRIAL: NCT03975816
Title: Changhua Christian Hospital, Department of Anesthesiology
Brief Title: The Application of Analgesia Nociception Index as an Objective Labor Pain Assessment During Epidural Analgesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ANIpainlesslabor
Record Dates: First submitted 2019-04-18; First posted 2019-06-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Labor Pain
Keywords: Analgesia nociception index; Painless labor; epidural analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Analgesia nociception index — Monitor the maternity with Analgesia nociception index

SUMMARY:
Epidural analgesia is considered an effective and safe method for obstetric pain control. Currently, self-assessment pain scales remain to be the gold standard in labor pain evaluation after the administration of epidural analgesia. However, individual patient susceptibility to pain perception makes difficulties for the clinicians to assess the effectiveness of painless labor precisely. The aim of this study is to evaluate the validity of ANI in obstetric pain monitoring during epidural analgesia.

DETAILED DESCRIPTION:
Epidural analgesia is considered an effective and safe method for obstetric pain control. Currently, self-assessment pain scales remain to be the gold standard in labor pain evaluation after the administration of epidural analgesia. However, individual patient susceptibility to pain perception makes difficulties for the clinicians to assess the effectiveness of painless labor precisely. Without a convincing objective tool for obstetric pain evaluation during epidural analgesia, the clinicians are hard to adjust adequate epidural drug dosage. Establishing an objective pain index would help the clinicians to have a better pain management during labor.

In 2012, M. Le Guen et al. demonstrated a linear relationship between visual analogical pain scores(VAS) and Analgesia Nociception Index (ANI) values during labor. Their efforts started the application of ANI in obstetric pain monitoring. However, the reliability of ANI in obstetric pain monitoring under epidural analgesia have not yet been verified. The aim of this study is to evaluate the validity of ANI in obstetric pain monitoring during epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with gestational age more than 35 weeks
* Ages between 20 to 50
* Received epidural analgesia
* American Society of Anesthesiologists classification I or II.

Exclusion Criteria:

* 1. Who refused to join the study
* 2. With a history of arrhythmia
* 3. American Society of Anesthesiologists (ASA)Classification >= III
* 4. With a history of cardiovascular, pulmonary, endocrine, neurologic or psychiatric disease
* 5.Using medications that affecting heart rate
* 6. Cannot understand the explanation of the study
* 7. High-risk gestation
* 8. Known fetal anomaly

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturients received epidural analgesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-17 (Actual); Primary Completion 2022-08-21 (Estimated); Study Completion 2023-08-21 (Estimated)

PRIMARY OUTCOMES:
The correlation of subjective pain measurement by the VAS score and objective pain measurement by the ANI(Analgesia Nociception Index) score | 90 minutes
  The VAS(visual analog scale) score is a subjective measure for pain. Scores are recorded by making a handwritten mark by the patient on a 10-cm line that represents a continuum between "no pain" and "worst pain." The score will be transferred to a 0-100 index by divided 10 with the distance from the starting point to the written mark (in centimeter) and multiplied by 100. The ANI (Analgesia Nociception Index) score is a 0-100 index derived from heart rate variability which was applied as an objective pain measurement. The larger the index indicated less pain. The correlation of the VAS score and the ANI score will be analyzed to verified the strength of the ANI score in evaluating labor pain during epidural analgesia.

SECONDARY OUTCOMES:
The correlation of uterine contraction strength measured by cardiotocography and the ANI (Analgesia Nociception Index) score | 90 Minutes
  Uterine contraction strength was measured by external cardiotocography with a scare from 0-100.The ANI (Analgesia Nociception Index) score is a 0-100 index derived from heart rate variability which was applied as an objective pain measurement. The larger the index indicated less pain. The correlation of the uterine contraction strength and the ANI score will be analyzed to verified if the ANI score changing with related to uterine contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Lun Tsao, MD, Study Director — Changhua Christian Hospital, Department of Anesthesiology
Locations (1):
- Changhua Christian hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individuals participants data for primary outcome measure will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available within 1 year of study completion
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Le Guen M, Jeanne M, Sievert K, Al Moubarik M, Chazot T, Laloe PA, Dreyfus JF, Fischler M. The Analgesia Nociception Index: a pilot study to evaluation of a new pain parameter during labor. Int J Obstet Anesth. 2012 Apr;21(2):146-51. doi: 10.1016/j.ijoa.2012.01.001. Epub 2012 Feb 21. PMID 22360936